CLINICAL TRIAL: NCT00326833
Title: How Many Patients Are in Need of Vitamin B12 Injections?
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Anne-Mette Hvas, Aarhus University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2005-0198
Record Dates: First submitted 2006-05-16; First posted 2006-05-17 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 2008-08

CONDITIONS: Vitamin B12 Deficiency
Keywords: Vitamin B12 deficiency; Vitamin B12 absorption; Holotranscobalamin
MeSH Terms: conditions — Vitamin B 12 Deficiency | interventions — Vitamin B 12

INTERVENTIONS:
Drug: vitamin B12 — 9 µg vitamin B12 three times daily for two days (CobaSorb)

SUMMARY:
The clinical consequences of vitamin B12 deficiency include megaloblastic anemia and neurological disorders. Therefore, a proper and timely diagnosis and treatment is important. The use of sensitive biochemical markers such as methylmalonic acid for the diagnosis of vitamin B12 deficiency have increased since the 1980s. Consequently, the number of individuals treated with vitamin B12 has increased significantly.

The objective of this project is to study the actual need for vitamin B12 injections in the group of individuals who have already started treatment. In order to investigate this, the investigators stop vitamin B12 treatment in this group, and look for signs of vitamin B12 deficiency by monitoring changes in biochemical and hematological markers. Furthermore, they will test if the individuals are able to absorb a physiological dose of vitamin B12 using a recently developed absorption test (CobaSorb). If a physiological dose can be absorbed, the vitamin B12 injections can be replaced with tablets. In the end, the investigators hope to be able to divide the patients into three groups:

1. need life long injections with vitamin B12,
2. only need supplementations with a small dose of oral vitamin B12, and
3. no need for further vitamin B12 treatment.

The perspective is that the new information from this study might be used for a future strategy for vitamin B12 treatment.

DETAILED DESCRIPTION:
The clinical consequences of vitamin B12 deficiency include megaloblastic anemia and neurological disorders. Therefore, a proper and timely diagnosis and treatment is important. The use of sensitive biochemical markers such as methylmalonic acid for the diagnosis of vitamin B12 deficiency have increased since the 1980s. Consequently, the number of individuals treated with vitamin B12 has increased significantly.

The objective of this project is to study the actual need for vitamin B12 injections in the group of individuals who have already started treatment. In order to investigate this, the investigators stop vitamin B12 treatment in this group, and look for signs of vitamin B12 deficiency by monitoring changes in biochemical and hematological markers. Furthermore, they will test if the individuals are able to absorb a physiological dose of vitamin B12 using a recently developed absorption test (CobaSorb). If a physiological dose can be absorbed, the vitamin B12 injections can be replaced with tablets. In the end, the investigators hope to be able to divide the patients into three groups:

1. need life long injections with vitamin B12,
2. only need supplementations with a small dose of oral vitamin B12, and
3. no need for further vitamin B12 treatment.

The perspective is that the new information from this study might be used for a future strategy for vitamin B12 treatment.

ELIGIBILITY:
Inclusion Criteria:

* Above 17 years old
* Have received vitamin B12 treatment for at least one year
* Capable of reading and understanding Danish

Exclusion Criteria:

* Pregnant or nursing women
* Not capable of giving informed consent
* Acute infection during the 3-day examination of vitamin B12 absorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-01; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Change in plasma cobalamins | Every month
Change in plasma methylmalonic acid | Every month
Change in plasma holotranscobalamin | Every month

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Mette Hvas, MD, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Anne-Mette Hvas, Aarhus N, Denmark

REFERENCES:
- [Derived] Hvas AM, Morkbak AL, Hardlei TF, Nexo E. The vitamin B12 absorption test, CobaSorb, identifies patients not requiring vitamin B12 injection therapy. Scand J Clin Lab Invest. 2011 Sep;71(5):432-8. doi: 10.3109/00365513.2011.581389. Epub 2011 May 30. PMID 21623649